CLINICAL TRIAL: NCT00000637
Title: A Randomized Comparative Trial of Zidovudine (AZT) Versus 2',3'-Dideoxyinosine (ddI) Versus AZT Plus ddI in Symptomatic HIV-Infected Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 152; 11127 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To compare the effectiveness of treatment with zidovudine (AZT) compared to didanosine (ddI) and compared to the combination of AZT and ddI as determined by survival and disease progression. To compare the relative safety and tolerance of AZT versus ddI versus AZT plus ddI in symptomatic HIV infected children; to compare the virological and immunological parameters in the three treatment groups. AZT has been shown to delay the progression of AIDS in HIV infected individuals. However, bone marrow toxicity is a frequent adverse effect. Also, HIV resistance to AZT sometimes occurs in patients who initially respond to treatment, but later have progression of the disease. Thus, new drug treatments are needed. Studies of ddI in adults and children indicate some effectiveness of the drug. A direct comparison of AZT and ddI treatment in children has not been made. Combination antiviral treatment (AZT plus ddI) may give added therapeutic benefit to children.

DETAILED DESCRIPTION:
AZT has been shown to delay the progression of AIDS in HIV infected individuals. However, bone marrow toxicity is a frequent adverse effect. Also, HIV resistance to AZT sometimes occurs in patients who initially respond to treatment, but later have progression of the disease. Thus, new drug treatments are needed. Studies of ddI in adults and children indicate some effectiveness of the drug. A direct comparison of AZT and ddI treatment in children has not been made. Combination antiviral treatment (AZT plus ddI) may give added therapeutic benefit to children.

Patients are placed by random selection into one of three groups to receive either AZT alone, ddI alone, or AZT and ddI. This is a double-blind study: neither patient nor treating physician knows which group patient is in. If patients are receiving either AZT or ddI alone and they develop drug toxicity (after dose reduction), or if HIV disease progresses, the alternative single drug is offered. If patients receiving both drugs develop drug toxicity (despite dose reduction) or if HIV disease progresses, they discontinue study drug and are offered the best alternative therapy. PER AMENDMENT 6/26/95: Initial monotherapy AZT arm is unblinded and no further crossover therapy for any arm is permitted. Patients who reach crossover criteria on initial blinded ddI or AZT+ddI will be unblinded and permanently discontinued from study drugs.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acetaminophen, ibuprofen, or aspirin, but not on a continual basis for > 72 hours.
* Systemic ketoconazole and fluconazole for acute therapy.

Recommended:

* Prophylaxis for PCP. (Primary prophylaxis with TMP / SMX is encouraged.) IV pentamidine may be used in selected cases if not administered on a weekly basis.

Patients must have the following:

* HIV infection.
* Children randomized prior to their eighteenth birthday are eligible. Co-enrollment in either ACTG 179 or 189 is permitted.

Prior Medication:

Allowed:

* Up to six weeks of antiretroviral or immunomodulator treatment excluding steroids and intravenous immunoglobulin.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active malignancy.
* Pancreatitis or history of pancreatitis within one year prior to study entry associated with compatible symptoms.
* History of uncontrolled seizure disorder.
* Grade 3 or higher peripheral neuropathy.
* Cardiomyopathy.

Concurrent Medication:

Excluded:

* Chemotherapy for malignancy.
* Oral acidifying agents.
* Acetaminophen, ibuprofen, or aspirin on a continual basis for > 72 hours.
* Ketoconazole or fluconazole for prophylaxis.
* Drugs with potential to cause peripheral neuropathy or pancreatitis should not be given daily for > 4 weeks.

Patients with the following are excluded:

* Active malignancy.
* Pancreatitis or history of pancreatitis within one year prior to study entry associated with compatible symptoms.
* History of uncontrolled seizure disorder.
* Grade 3 or higher peripheral neuropathy.

Prior Medication:

Excluded:

* Steroids.
* Intravenous immunoglobulin.
* Antiretroviral drugs or specific immunomodulator treatment (excluding steroids and intravenous immunoglobulin) for > 6 weeks and within 7 days prior to study entry.

Prior Treatment:

Excluded:

* Red blood cell transfusion within four weeks prior to study entry.

Ongoing drug or alcohol use.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 819
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baker C, Study Chair; Englund J, Study Chair
Locations (80):
- United States (76):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - Kaiser Permanente / UCLA Med Ctr, Downey, California
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - Huntington Memorial Hosp / Children's Hosp of Los Angeles, Pasadena, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Stanford Univ School of Medicine / Pediatrics, Stanford, California
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Connecticut Health Ctr, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - St Louis Univ School of Medicine, St Louis, Missouri
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Robert Wood Johnson Med School / Hershey Med Ctr, New Brunswick, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - King's County Hosp Ctr / Pediatrics, Brooklyn, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - SUNY / Health Sciences Ctr at Brooklyn / Pediatrics, Brooklyn, New York
  - Children's Hosp Pact Prog / Children's Hosp of Buffalo, Buffalo, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Lincoln Hosp Ctr, The Bronx, New York
  - Bronx Lebanon Hosp Ctr / Pediatrics, The Bronx, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Westchester Hosp, Valhalla, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Cincinnati Children's Hosp / Univ Hosp, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Hemophilia Ctr of Western PA / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hosp / Brown Univ, Providence, Rhode Island
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of Seattle, Seattle, Washington
- Puerto Rico (4):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - UPR Children's Hosp / UPR School of Medicine, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Raskino C, Pearson DA, Baker CJ, Lifschitz MH, O'Donnell K, Mintz M, Nozyce M, Brouwers P, McKinney RE, Jimenez E, Englund JA. Neurologic, neurocognitive, and brain growth outcomes in human immunodeficiency virus-infected children receiving different nucleoside antiretroviral regimens. Pediatric AIDS Clinical Trials Group 152 Study Team. Pediatrics. 1999 Sep;104(3):e32. doi: 10.1542/peds.104.3.e32. PMID 10469815
- [Background] Grubman S. Pediatric treatment update. GMHC Treat Issues. 1996 Mar;10(3):7-9. PMID 11363392
- [Background] Glick ME. CTG studies yield results. AIDS Clinical Trials Group. NIAID AIDS Agenda. 1995 Spring:8-9. PMID 11362451
- [Background] Rogers MF, Mofenson LM, Moseley RR. Reducing the risk of perinatal HIV transmission through zidovudine therapy: treatment recommendations and implications. J Am Med Womens Assoc (1972). 1995 May-Aug;50(3-4):78-82, 93. PMID 7657952
- [Background] Nielsen K, Wei LS, Sim MS, Deveikis A, Keller M, Stiehm ER, Frenkel LM, Bryson YJ. Correlation of clinical progression in human immunodeficiency virus-infected children with in vitro zidovudine resistance measured by a direct quantitative peripheral blood lymphocyte assay. J Infect Dis. 1995 Aug;172(2):359-64. doi: 10.1093/infdis/172.2.359. PMID 7622878
- [Background] Palumbo PE, Raskino C, Fiscus S, Pahwa S, Fowler MG, Spector SA, Englund JA, Baker CJ. Predictive value of quantitative plasma HIV RNA and CD4+ lymphocyte count in HIV-infected infants and children. JAMA. 1998 Mar 11;279(10):756-61. doi: 10.1001/jama.279.10.756. PMID 9508151
- [Background] McKinney RE Jr, Wilfert C. Growth as a prognostic indicator in children with human immunodeficiency virus infection treated with zidovudine. AIDS Clinical Trials Group Protocol 043 Study Group. J Pediatr. 1994 Nov;125(5 Pt 1):728-33. doi: 10.1016/s0022-3476(94)70065-6. PMID 7965424
- [Background] James JS. AZT, ddI, and ddC combinations at FDA advisory hearing. Food and Drug Administration. AIDS Treat News. 1996 Apr 5;(no 244):6. PMID 11363307
- [Background] Englund JA, Baker CJ, McKinney RE, Raskino CL, Fowler MG, Lifschitz MC. Results of ACTG 152, a randomized comparative trial of zidovudine (ZDV), didanosine (ddI), and ZDV/ddI combination therapy in symptomatic HIV-infected children. Program Abstr Intersci Conf Antimicrob Agents Chemother. 1996 Sep 15-18:213 (abstract no I150)
- [Background] Englund JA, Baker CJ, Raskino C, McKinney RE, Petrie B, Fowler MG, Pearson D, Gershon A, McSherry GD, Abrams EJ, Schliozberg J, Sullivan JL. Zidovudine, didanosine, or both as the initial treatment for symptomatic HIV-infected children. AIDS Clinical Trials Group (ACTG) Study 152 Team. N Engl J Med. 1997 Jun 12;336(24):1704-12. doi: 10.1056/NEJM199706123362403. PMID 9182213
- [Background] Capparelli EV, Englund JA, Connor JD, Spector SA, McKinney RE, Palumbo P, Baker CJ. Population pharmacokinetics and pharmacodynamics of zidovudine in HIV-infected infants and children. J Clin Pharmacol. 2003 Feb;43(2):133-40. doi: 10.1177/0091270002239821. PMID 12616665
- [Background] Chantry CJ, Byrd RS, Englund JA, Baker CJ, McKinney RE Jr; Pediatric AIDS Clinical Trials Group Protocol 152 Study Team. Growth, survival and viral load in symptomatic childhood human immunodeficiency virus infection. Pediatr Infect Dis J. 2003 Dec;22(12):1033-9. doi: 10.1097/01.inf.0000100575.64298.bc. PMID 14688560